CLINICAL TRIAL: NCT04073953
Title: Metabolism and Pharmacokinetics of Primaquine Enantiomers in G6PD Deficient Human Volunteers Receiving a Five Day Dose Regimen
Brief Title: Primaquine Enantiomers in G6PD Deficient Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PQ Study 3
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: G6PD Deficiency
Keywords: G6PD; Hemolysis; Primaquine; Pharmacokinetics; Malaria
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency; Hemolysis; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RPQ (-) enantiomer (Experimental): Cohort 1 will receive 15mg of RPQ every day for 5 days. Cohort 2 will receive 22.5 mg of RPQ every day for five days.
  Interventions: Drug: RPQ
- SPQ (+) enantiomer (Experimental): Cohort 1 will receive 15mg of SPQ every day for 5 days. Cohort 2 will receive 22.5 mg of SPQ every day for five days.
  Interventions: Drug: SPQ
- Placebo (Placebo Comparator): Cohort 1 will receive placebo capsules every day for 5 days. Cohort 2 will receive placebo capsules every day for five days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPQ — The study will compare the individual enantiomers of Primaquine -R-(-)-PQ, S-(+)-PQ, and Placebo.
  Other Names: R-(-) Enantiomer of Primiquine Phosphate
  Arms: RPQ (-) enantiomer
Drug: SPQ — The study will compare the individual enantiomers of Primaquine -R-(-)-PQ, S-(+)-PQ, and Placebo.
  Other Names: S-(+) Enantiomer of Primaquine Phosphate
  Arms: SPQ (+) enantiomer
Drug: Placebo — The study will compare the individual enantiomers of Primaquine -R-(-)-PQ, S-(+)-PQ, and Placebo.
  Arms: Placebo

SUMMARY:
This study is a single center, prospective, cross-over phase 1 trial. Eighteen subjects will be enrolled in the study evaluating the metabolism, pharmacokinetic behavior and tolerability of primaquine enantiomers and placebo over the course of 5 days.

DETAILED DESCRIPTION:
Each subject will receive a 15 mg dose of one enantiomer (SPQ or RPQ or Placebo) daily for up to 5 days, with careful monitoring of hematological parameters before and after each dose. In addition to the general CMP14 safety criteria, any subject who displays a fractional hemoglobin drop of 15% below his/her baseline value, then drug administration will stop (e.g. for baseline Hgb of 14 g/dL, if there is at any point a decrease of 2.1 g/dL). Hematocrit will be similarly monitored, with proportional stop criteria. Elevation in total bilirubin to 2.0 mg/dL or greater will also be used as a stopping criterion. After stopping drug administration (5 days or whenever stop criteria are met), subjects will have a 3-week washout period, and the study repeated with the other enantiomer, and similarly with Placebo.

ELIGIBILITY:
Inclusion Criteria:

* G6PD deficient, otherwise normal healthy adults aged 18 to 65

Exclusion Criteria:

* Known history of liver, kidney or hematological disease (other than G6PD deficiency)
* Known history of cardiac disease, non-sinus rhythm arrhythmia or QT prolongation
* Autoimmune disorders
* Report of an active infection
* Subject is pregnant or breast-feeding, or is expecting to conceive during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Methemoglobin concentration in blood from baseline | Days 0, 3, 5
  Change in Methemoglobin concentration in blood from baseline (% hemoglobin)

SECONDARY OUTCOMES:
Primaquine Plasma Concentration, ng/mL | Days 0, 3, 5
  Plasma concentrations of parent drug
Carboxy-Primaquine Plasma Contration, ng/mL | Days 0, 3, 5
  Plasma concentrations of carboxy-primaquine metabolite
Primaquine N-carbamoyl-glucuronide Plasma contration, ng/mL | Days 0, 3, 5
  Plasma concentrations of Primaquine N-carbamoyl-glucuronide metabolite
Primaquine Orthoquinone Plasma concentration, ng/mL | Days 0, 3, 5
  Plasma concentrations of Primaquine Orthoquinone metabolite
Change in Hematocrit (%) compared to baseline | Days 0, 3, 5
  Change in Hematocrit (%) compared to baseline
Change in Hemoglobin (g/dL) compared to baseline | Days 0, 3, 5
  Change in Hemoglobin (g/dL) compared to baseline
Change is AST (U/L) compared to baseline | Days 0, 3, 5
  Change is AST (U/L) compared to baseline; used to monitor liver function
Change in ALT (U/L) compared to baseline | Days 0, 3, 5
  Change in ALT (U/L) compared to baseline; used to monitor liver function
Change in total Bilirubin (mg/dL) compared to baseline | Days 0, 3, 5
  Change in total Bilirubin (mg/dL) compared to baseline; used to monitor liver function and red cell integrity

CONTACTS AND LOCATIONS:
Overall Officials: Larry Walker, Ph.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi, University, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No